CLINICAL TRIAL: NCT03564431
Title: The Study of Structural and Functional Brain Abnormalities and the Association With the Genetic Polymorphism in the Type 2 Diabetes Patient With Depression
Brief Title: The Imaging Genetic Study of Type 2 Diabetes and Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuqi Cheng, associate professor, Kunming Medical University
Other Study IDs: 841026
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: T2DM
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — perapheral blood DNA of all participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- controls
  Interventions: Device: Magnetic resonance
- T2DM patients
  Interventions: Device: Magnetic resonance
- depression patients
  Interventions: Device: Magnetic resonance
- T2DM with depression patients
  Interventions: Device: Magnetic resonance

INTERVENTIONS:
Device: Magnetic resonance — magnetic resonance spectrum of brain

SUMMARY:
To investigate the structural/functional abnormalities and the possible genetic endophenotypes of in the Type 2 Diabetes Patient With Depression.

DETAILED DESCRIPTION:
Diabetes and depression are harmful to human health,but they often co-exist.At present, the pathophysiological mechanisms underlying the comorbidity of diabetes and depression are discussed, including hypothalamic-pituitary-adrenal axis dysfunction, inflammation, epigenetics, disturbed circadian rhythms, environmental and behavioral factors,neuroimaging,etc.the purpose of the investigator's study is to investigate the structural/functional abnormalities and the possible genetic endophenotypes of in the Type 2 Diabetes Patient With Depression.

ELIGIBILITY:
Inclusion Criteria:

conform to type 2 diabetes, depression, diagnostic criteria of unrelated normal controls the han nationality patients; Aged 30 to 70 years of age, gender not limited; The patient or legal guardian have signed informed consent of patients.

Exclusion Criteria:

Magnetic resonance imaging has the contraindication, such as metal implants, claustrophobic, etc.

With severe body diseases, including inflammatory diseases and autoimmune diseases; Current or past history of nervous system disease or brain injury. Merge other severe mental illness or existing psychotic symptoms; Always have a mania, hypomania attack; Has a history of substance abuse; Pregnant women and nursing mothers; Estimated compliance is poorer, not partners; Is being treated for a mental drug therapy, and ECT, TMS; Patients with a body mass index > 35; There are currently no taking corticosteroids, immune regulator, etc. Now or ever did not suffer from patients with other diagnosis to the dsm-iv axis I; Merge the endocrine system disease, thyroid, adrenal gland and pituitary gland diseases, etc.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM and depression patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
the neuroimaging of Type 2 Diabetes and Depression | from 2017-12 to 2019-12
  the structure and function of Abnormalities in the T2DM Patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Xu, MD, Principal Investigator — Psychiatry department of KMU
Locations (1):
- Psychiatry department, The 1st Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui F, Ouyang ZQ, Zeng YZ, Ling BB, Shi L, Zhu Y, Gu HY, Jiang WL, Zhou T, Sun XJ, Han D, Lu Y. Effects of hypertension on subcortical nucleus morphological alternations in patients with type 2 diabetes. Front Endocrinol (Lausanne). 2023 Sep 13;14:1201281. doi: 10.3389/fendo.2023.1201281. eCollection 2023. PMID 37780620